CLINICAL TRIAL: NCT06708936
Title: A Single-arm, Open-label, Single-center, Multiple-dose Early Exploratory Clinical Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of KSD-201 in Patients With Advanced Clear Cell Renal Cell Carcinoma
Brief Title: KSD-201 Treatment for Advanced Clear Cell Renal Cell Carcinoma: an Early Exploratory Clinical Study
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Kousai Bio Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSD-201-CR001
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2024-11

CONDITIONS: Clear Cell Renal Cell Carcinoma (ccRCC)
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- KSD-201 (Experimental): Biological: Dendritic Cell Vaccine.Autologous monocyte-derived DCs pulsed with clear cell renal cell carcinoma-associated antigen.
  Interventions: Biological: KSD-201

INTERVENTIONS:
Biological: KSD-201 — Patients will receive approximately 5x10^6 cells/dose DC vaccine via subcutaneous injections bi-weekly,total 3-5 times.

SUMMARY:
The main purpse of this study is to evaluate the safety and tolerability of KSD-101 in patients with advanced clear cell renal cell carcinoma, to evaluate the initial clinical outcomes , immune response, and to evaluate the impact of KSD-201 on the quality of life in patients with advanced clear cell renal cell carcinoma.

DETAILED DESCRIPTION:
This study is a single-center, single-arm, open-label, dose-confirmation clinical trial designed to evaluate the safety, tolerability, immune response, and preliminary clinical efficacy of KSD-201 in the treatment of patients with advanced clear cell renal cell carcinoma. The study is conducted in two phases: the first phase is for dose-limiting toxicity (DLT) observation and dose confirmation; the second phase is an expansion study, where the investigators may add 3 to 6 subjects based on the safety and efficacy signals obtained from the first phase.

Enrolled subjects will undergo peripheral blood mononuclear cell collection. The collected material is transported via cold chain logistics to the dendritic cell vaccine preparation site, where the dendritic cell vaccine (KSD-201) is prepared using the subject's own monocytes. Once KSD-201 is successfully prepared, subjects will return to the hospital for KSD-201 injection according to the following method.

1. KSD-201 treatment dose: The provisional dosing is set at 5.0 × 10^6 cells/dose.
2. KSD-201 treatment frequency: a total of 3-5 times. The 4th and 5th times are booster treatments, which need to be decided by the investigator according to the condition of the subjects.
3. Dosing interval: 2 weeks. The interval may be adjusted based on the subject's condition during the intensive treatment phase.
4. KSD-201 route of administration: subcutaneous injection.
5. Administration site: near the axillary lymph node or inguinal lymph node.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects and/or their legal guardians agree to participate and sign the ICF. 2. Male or female subjects aged 18 years and above on the day of ICF signing. 3. Patients with advanced clear cell renal cell carcinoma, confirmed by pathological tissue examination, who have failed standard therapy (failure of standard therapy refers to disease progression confirmed by imaging during or after at least one systemic regimen, or intolerance to such regimen, which includes tyrosine kinase inhibitors such as sunitinib, axitinib, pazopanib, sorafenib, among others, as well as everolimus and immune checkpoint inhibitors), and for whom no effective treatment measures are available, with the condition posing a serious threat to their lives.

  4. According to RECIST v1.1 criteria, there should be at least one measurable lesion.

  5. Eastern Cooperative Oncology Group (ECOG) score of 0-1. 6. Eligible for leukapheresis and has no other contraindications for cell collection.

  7. Must have adequate organ function：
  * Hematology test: Monocyte count ≥ 0.1 × 10^9/L, neutrophil count ≥ 1.5 × 10^9/L, hemoglobin ≥ 90 g/L, platelet count ≥ 100 × 10^9/L， and no blood transfusion or blood products within 28 days prior to leukapheresis, and no use of hematopoietic growth factors or other drugs to correct blood cells.
  * Liver function: ALT, AST ≤ 2.5 × ULN and TBIL ≤ 1.5 × ULN [for patients with liver metastases: ALT, AST ≤ 5 × ULN and TBIL ≤ 2 × ULN]
  * Kidney function: Creatinine ≤ 1.5 × ULN
  * Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 50%
  * pulmonary function：Pulse oximetry saturation ≥ 94%.
  * Coagulation function: Fibrinogen ≥ 1.0 g/L, activated partial thromboplastin time (APTT) ≤ 1.5 × ULN, prothrombin time (PT) ≤ 1.5 × ULN 8. Patient's corresponding lymph node regions meet the requirements for subcutaneous injection.

    9. Male and female subjects of reproductive age agree to take non-pharmacological contraceptive measures from signing the ICF until 6 months after the last dose.

Exclusion Criteria:

* 1. Within 4 weeks prior to apheresis, patients have received any chemotherapy, immunosuppressive drugs, or other medicinal treatments, or have undergone less than 5 drug half-lives (whichever is shorter), and within 2 weeks prior to apheresis, they have undergone systemic radiation therapy.

  2. Underwent allogeneic transplantation prior to enrollment. 3. Received (attenuated) live vaccines within 4 weeks prior to enrollment. 4. Participated in other clinical studies within 4 weeks prior to enrollment and received at least one dose of the investigational product.

  5. Underwent therapeutic surgery within 4 weeks prior to enrollment, or plan to undergo major surgery during the study, except diagnostic, biopsy and drainage procedures.

  6. Presence of uncontrolled infectious disease within 4 weeks prior to enrollment.

  7. Receiving systemic corticosteroid therapy prior to screening and require long-term systemic corticosteroids during the treatment period (except inhalation or topical application) as judged by the investigator, or received systemic corticosteroid therapy (except inhalation or topical application) within 72 hours prior to administration.

  8. Active central nervous system metastases/lesions (e.g., brain edema requiring hormone intervention or brain metastases).

  9. Severe cardiovascular diseases:
  * Grade ≥ 3 cardiovascular diseases according to the New York Heart Association (NYHA) classification within 6 months prior to enrollment.
  * Unstable angina or severe arrhythmias requiring medication.
  * Other significant ECG abnormalities, including second-degree type 2 atrioventricular block, third-degree atrioventricular block, bradycardia (ventricular rate < 50 beats/min with clinical symptoms), etc.

    10. Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and increased peripheral blood hepatitis B virus (HBV) DNA titer above the ULN; positive for hepatitis C virus (HCV) antibody and peripheral blood HCV RNA; positive for human immunodeficiency virus (HIV) antibody; positive for syphilis-specific antibodies.

    11. Have not recovered to normal or Grade ≤ 1 from prior treatment-induced AEs prior to enrollment, except alopecia (any grade) and peripheral neuropathy (Grade ≤ 2).

    12. Other active malignancies within the past 3 years, except for curable cancers that have been markedly cured, such as basal or squamous cell carcinoma, cervical or breast cancer in situ.

    13. Prior history of severe drug allergies or history of penicillin allergy. 14. Substance abuse/addiction. 15. Women who are pregnant or nursing. 16. Other serious medical conditions, including liver disease, kidney disease, neurological/psychiatric disorders, endocrine disorders, hematologic disorders, and immune system disorders, which will render a subject unsuitable for participation in the study as judged by the investigator.

    17. Other conditions that render a subject unsuitable for enrollment as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
DLT | From the infusion (Day 0) to Day 28
  Incidence and number of dose-limiting toxicities
Safety | 1 year after DC Vaccines injection
  Incidence and severity of AEs, including vital signs, physical examination, and laboratory tests

SECONDARY OUTCOMES:
Objective response rate (ORR) | 1 year after DC Vaccines injection
  The percentage of participants who achieved PR or better response
Disease control rate (DCR) | 1 year after DC Vaccines injection
  The percentage of participants who achieved SD or better response
Duration of response (DOR) | 1 year after DC Vaccines injection
  DOR will be calculated among responders (with a PR or better response) from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease
Progression-free survival (PFS) | 1 year after DC Vaccines injection
  The time from the start of CAR-GPRC5D treatment for the participants to the first time of disease progression or death for any reason
Overall survival (OS) | 1 year after DC Vaccines injection
  OS is measured from the date of the initial injection of DC Vaccines to the date of the participant's death
Levels of various lymphocyte subsets | 1 year after DC Vaccines injection
  total T lymphocytes, activated T lymphocytes, helper T lymphocytes, cytotoxic T lymphocytes, regulatory T lymphocytes, total B lymphocytes and total NK cells in peripheral blood will be assessed to monitor changes
EQ-5D-5L | Up to 1 year
  The change from baseline in scores of EQ-5D-5L endpoints will be analyzed by age group or indication group
QLQ-C30 | Up to 1 year
  The change from baseline in scores of QLQ-C30 endpoints will be analyzed by age group or indication group

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided